CLINICAL TRIAL: NCT05888636
Title: Transcriptomics and Epigenetics Analysis for Biomarkers Identification Involved in Drug-resistance Mechanisms of Multiple Myeloma
Brief Title: Transcriptomics and Epigenetics Analysis in Drug-Resistance of Multiple Myeloma
Acronym: TEDROMM
Status: Recruiting | Type: Observational
Sponsor: Regina Elena Cancer Institute (Other)
Collaborators: Campus Bio-Medico University (Other); University of Rome Tor Vergata (Other); S.Eugenio Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RS1237
Record Dates: First submitted 2023-03-24; First posted 2023-06-05 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Chromatin Immunoprecipitation Sequencing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- MGUS
  Interventions: Other: ChIP-seq, NGS, ATAC-seq
- MM smouldering
  Interventions: Other: ChIP-seq, NGS, ATAC-seq
- Syntomatic MM
  Interventions: Other: ChIP-seq, NGS, ATAC-seq

INTERVENTIONS:
Other: ChIP-seq, NGS, ATAC-seq — Bone narrow sampling

SUMMARY:
Multiple Myeloma (MM) is the more common hematological neoplastic disease second only to Hodgkin lymphoma. In MM patients, mutated genes are mainly KRAS (23%), NRAS (20%), FAM46C (11%), DIS3 (11%) e TP53 (8%). Epigenetics studies suggested that Changes in histone modifications and DNA methylation pattern, as well as non-coding RNAs (miRNAs) expression are involved in MM development. In particular, it has been shown that the aberrant expression of different miRNAs could discriminate healthy from ill patients. Unfortunately, the main critical issue for an effective treatment of MM is the intrinsic or acquired resistance to pharmacological treatments, due also to a plasmacellular clonal heterogeneity.

The prospective study will involve a patient cohort with MGUS, MM smouldering and MM, with the aim to characterize different transcriptional and epigenetic features, also including miRNAs, among MM cells susceptible or resistant to conventional therapies. The final goal is to identify new prognostic and predictive biomarkers that could be used as therapeutic tools to improve clinical targeted therapies.

ELIGIBILITY:
Inclusion Criteria:

- Compare Transcriptomics and epigenetic profile

Exclusion Criteria:

* No exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: For the study, samples from patients with MGUS, MM smouldering and syntomatic MM will be used
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-06-18 (Actual); Primary Completion 2023-11-11 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Transcriptomics variations in treated and non-treated MGUS, MM smouldering and syntomatic MM samples | 12 months
  Characterize genetic/epigenetic profile of cells resistant to the treatment sampled from MM patients before and after treatement.
Epigenetics variations in treated and non-treated MGUS, MM smouldering and syntomatic MM samples | 12 months
  Quantify genetic/epigenetic profile of cells resistant to the treatment sampled from MM patients before and after treatement.

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Fanciulli, PhD, Principal Investigator — IRCCS "Regina Elena" National Cancer Institute
Locations (2):
- Italy (2):
  - Regina elena Cancer Institute, Roma
  - "Regina Elena" National Cancer Institute, Rome

IPD SHARING:
Plan to Share IPD: Undecided